CLINICAL TRIAL: NCT00800397
Title: Evaluation of the Noga System: Detecting of Respiratory Related Sleep Disorders in Cardiac Patients
Status: Completed | Type: Observational
Sponsor: WideMed LTD. (Industry)
Responsible Party: Anya Eldan, WideMed LTD.
Other Study IDs: MorpheusHx002
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Medical literature has shown that 1 out of 2 patients that are admitted to the hospital as a cardiac patient, will be found suffering from sleep breathing disorders. The medical literature also shows that there is an advantage of treating the sleep breathing disorders in addition to treating the cardiac disease or evaluating the heart failure condition to provide better clinical outcomes.this study is evaluating the ability to detect sleep and cardiac related breathing disordered.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is hospitalized in the cardiology department or in the sleep lab.
2. Patients who is willing and able to tolerate a full night Polysomnography
3. Patient is not receiving oxygen treatment
4. Patients is 18 years of age or above
5. Patient is able and willing to sign the institution human subjects committee approved Informed Consent Form.

Exclusion Criteria:

1. Patients can not tolerate a full night Polysomnography.
2. Patient is receiving oxygen.
3. Participation in a clinical trial within the last 60 days and during the study.
4. Life expectancy < 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac and suspected sleep disordered breathing patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Detection of Cheyne Stokes respiration | over night

SECONDARY OUTCOMES:
Sleep and sleep apnea parameters | over night
AH>=15 | over night
plethysmography derived respiration signal | over night
Total duration of Cheyne Stokes | over night

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown memorial hospital, Morristown, New Jersey, United States